CLINICAL TRIAL: NCT04336540
Title: Socioeconomic Position and the Impact of Increasing Availability of Lower Energy Meals vs. Menu Energy Labelling on Food Choice in Virtual Full-service Restaurants: Two Randomized Control Trials
Brief Title: Increasing Availability of Lower Energy Meals vs. Menu Energy Labelling on Food Choice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Responsible Party: Principal Investigator, Eric Robinson, Principal Investigator, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 803194 1B2
Record Dates: First submitted 2020-04-02; First posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Nutrition Poor; Obesity; Diet, Healthy; Food Selection
MeSH Terms: conditions — Malnutrition; Obesity; Food Preferences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Energy labelling (Experimental): Energy labelling provided on restaurant menus
  Interventions: Other: Menu configuration (presence of energy labelling)
- No energy labelling (No Intervention): No energy labelling provided on restaurant menus
- Increased availability of lower energy meals (Experimental): Higher proportion of meals are 600kcals or less
  Interventions: Other: Menu configuration (presence of energy labelling); Other: Menu configuration (more lower energy options added)
- Baseline availability of lower energy meals (No Intervention): Proportion of meals that are 600kcals or less at baseline level

INTERVENTIONS:
Other: Menu configuration (presence of energy labelling) — Restaurant menus are altered to accommodate energy labelling intervention
  Arms: Energy labelling; Increased availability of lower energy meals
Other: Menu configuration (more lower energy options added) — Restaurant menus are altered to include more lower energy options
  Arms: Increased availability of lower energy meals

SUMMARY:
Two randomized control trials examining human food choice (i.e. selection of high energy 'unhealthy' foods vs. selection of healthier foods). Interventions: In a between-subjects design, participants (recruitment stratified by socioeconomic position) made food choices (main dish, plus optional sides and desserts) in the absence vs. presence of menu energy labelling and from menus with baseline (10%) vs. increased availability (50%) of lower energy main dishes. Main outcome measures: Average energy content (kcal) of main dish chosen and average total energy content of all food ordered, including optional sides and desserts.

DETAILED DESCRIPTION:
See attached protocol documents.

ELIGIBILITY:
Inclusion Criteria:

* Participants were eligible to participate if they were US residents, aged of 18 or above, fluent in English, had access to a computer with an internet connection and had no dietary restrictions

Exclusion Criteria:

* See above.

Stratification Criteria:

- We aimed to recruit a sample stratified by gender (approx. 50/50) and highest educational qualification (approx. 40% high school or less, 60% above high school) to be broadly representative of US adults.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2091 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Energy ordered from main menu | 15-20 minutes (the time frame denotes time taken to make the menu order and there is no follow up
  Total kcal content of main menu order

SECONDARY OUTCOMES:
Total energy ordered | 15-20 minutes (the time frame denotes time taken to make the menu order and there is no follow up
  Total kcal content of all food ordered (including sides, desserts)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Robinson, PhD, Principal Investigator — University of Liverpool
Locations (1):
- University of Liverpool, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Shared on the Open Science Framework
Supporting Information: Study Protocol, SAP
Time Frame: On publication, indefinitely
Access Criteria: Open website

REFERENCES:
- [Derived] Marty L, Reed SM, Jones AJ, Robinson E. Increasing availability of lower energy meals vs. energy labelling in virtual full-service restaurants: two randomized controlled trials in participants of higher and lower socioeconomic position. BMC Public Health. 2021 May 25;21(1):975. doi: 10.1186/s12889-021-11007-0. PMID 34034699

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT04336540/Prot_SAP_000.pdf